CLINICAL TRIAL: NCT01254344
Title: A Phase III, Randomized, Double-Blind, Active Comparator-Controlled Clinical Trial to Study the Efficacy and Safety of Ertapenem Sodium (MK-0826) Versus Ceftriaxone Sodium/Metronidazole for the Prophylaxis of Surgical Site Infection Following Elective Colorectal Surgery in Chinese Adults
Brief Title: Efficacy and Safety of Ertapenem Sodium (MK-0826) Following Colorectal Surgery in Chinese Adults (MK-0826-056)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0826-056
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Results first posted 2012-11-16 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Infection; Surgical Site Infection
Keywords: Colorectal surgery
MeSH Terms: conditions — Infections; Surgical Wound Infection | interventions — Ertapenem; L 749345; Ceftriaxone; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ertapenem sodium 1 g (Experimental): Ertapenem sodium 1 g administered intravenously (IV) as a single dose followed by matching placebo to metronidazole administered IV as a single dose
  Interventions: Drug: ertapenem sodium; Drug: placebo to metronidazole
- Ceftriaxone sodium 2 g (Active Comparator): Ceftriaxone sodium 2 g administered intravenously (IV) as a single dose followed by metronidazole 500 mg administered IV as a single dose
  Interventions: Drug: ceftriaxone sodium; Drug: metronidazole

INTERVENTIONS:
Drug: ertapenem sodium — Ertapenem sodium 1 g administered IV as a single dose over 30 minutes within 2 hours prior to the initial surgical incision
  Other Names: MK-0826; INVANZ®
  Arms: Ertapenem sodium 1 g
Drug: ceftriaxone sodium — Ceftriaxone sodium 2 g administered IV as a single dose over 30 minutes within 2 hours prior to the initial surgical incision
  Other Names: Rocephin®
  Arms: Ceftriaxone sodium 2 g
Drug: placebo to metronidazole — Placebo (0.9% sodium chloride) administered IV as a single dose over 30 minutes within 2 hours prior to the initial surgical incision
  Arms: Ertapenem sodium 1 g
Drug: metronidazole — Metronidazole 500 mg administered IV as a single dose over 30 minutes within 2 hours prior to the initial surgical incision
  Other Names: Flagyl®
  Arms: Ceftriaxone sodium 2 g

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ertapenem sodium compared with ceftriaxone sodium/metronidazole for the prophylaxis of surgical site infection following elective colorectal surgery in Chinese adults. This study is designed to demonstrate that ertapenem sodium is non-inferior to ceftriaxone sodium/metronidazole in this participant population.

ELIGIBILITY:
Inclusion Criteria:

- Participant is scheduled to undergo elective colon or colorectal surgery by

laparotomy that is scheduled in advance with adequate time prior to surgery to

complete preoperative bowel preparation.

- Participant is a Chinese adult between the ages of more than 18 years old and

less than 81 years old.

- Participant is highly unlikely to conceive.

Exclusion Criteria:

* Participant is undergoing emergency colon or colorectal surgery.
* Participant requires a second planned colorectal surgery or other surgery requiring antibiotic prophylaxis within the 4-week follow-up period.
* Participant is undergoing laparoscopic-assisted surgery.
* Participant is undergoing an isolated rectal procedure.
* Participant has a decompensated intestinal obstruction.
* Participant has active inflammatory bowel disease involving the colon (i.e.,

ulcerative colitis or Crohn's disease).

* Participant is scheduled to undergo an elective colorectal procedure for revision of a previous operation involving a large bowel resection.
* Participant has a bacterial infection at the time of surgery.
* Participant requires or is anticipated to need the administration of other (nonstudy therapy) systemic antimicrobial therapy within 1 week prior to surgery or at any time during this study.
* Participant is anticipated to receive either antibiotic or antiseptic peritoneal lavage during the surgery.
* Participant has a history of serious allergy, hypersensitivity (e.g., anaphylaxis), or any serious reaction to ertapenem sodium, ceftriaxone sodium, metronidazole, penicillin, or any cephalosporin, beta(β)-lactam, or nitroimidazole agents.
* Participant is breast feeding or plans to breast feed prior to the completion of the study period.
* Participant has neutropenia.
* Participant with immunosuppression due to an underlying disease, chronic

immunosuppressive therapy, or use of high-dose corticosteroids.

* Participant has a rapidly progressive or terminal illness.
* Participant is considered unlikely to survive through the expected 4-week study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Leng XS, Zhao YJ, Qiu HZ, Cao YK, Zhu WH, Shen JF, Paschke A, Dai WM, Caldwell N, Wang J. Ertapenem prophylaxis of surgical site infections in elective colorectal surgery in China: a multicentre, randomized, double-blind, active-controlled study. J Antimicrob Chemother. 2014 Dec;69(12):3379-86. doi: 10.1093/jac/dku302. Epub 2014 Aug 23. PMID 25151205

RESULTS

PARTICIPANT FLOW:
Groups:
- Ertapenem: Ertapenem sodium 1 g administered intravenously (IV) as a single dose followed by matching placebo to metronidazole administered IV as a single dose
- Ceftriaxone/Metronidazole: Ceftriaxone sodium 2 g administered intravenously (IV) as a single dose followed by metronidazole 500 mg administered IV as a single dose
Period: Overall Study
Arm/Group | Ertapenem | Ceftriaxone/Metronidazole
Started | 299 | 300
Treated | 290 | 297
Completed | 286 | 281
Not Completed | 13 | 19
Not completed — Adverse Event | 2 | 5
Not completed — Physician Decision | 7 | 4
Not completed — Protocol Violation | 1 | 4
Not completed — Withdrawal by Subject | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertapenem | Ceftriaxone/Metronidazole | Total
Number analyzed (Participants) | 290 | 297 | 587
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (11.4) | 59.1 (12.1) | 59.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 127 | 252
  Male | 165 | 170 | 335

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Success of Prophylaxis
Description: Percentage of participants who have no signs or symptoms of infection at the surgical site, do not require surgical intervention for infection, and have no need for further antimicrobial therapy
Time Frame: From study drug dose (day of surgery) up to 4 weeks post therapy
Population: Primary analysis results are for "evaluable-patients-only", defined as patients who received a complete dose of prophylaxis, underwent elective colorectal surgery with completion of bowel preparation procedure, had primary skin closure of the wound, and did not receive any prohibited systemic antibiotics or other prohibited anti-infective agents.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ertapenem | Ceftriaxone/Metronidazole
Number analyzed (Participants) | 251 | 248
percentage of participants | 90.4 [86.8 to 94.1] | 90.3 [86.6 to 94.0]
Statistical Analysis 1: Comparison: Ertapenem vs Ceftriaxone/Metronidazole; Test type: Non-Inferiority or Equivalence — Assuming a 70% rate (i.e., proportion of participants with "success of prophylaxis") for both groups and a significance level of 0.025, at least 200 evaluable participants per group were needed to have 90% probability that the lower limit of the 95% (two-sided) confidence interval for the difference in the response rates between the 2 groups was greater than -15 percentage points; Miettinen and Nurminen; Difference in percentage of prophylaxis = 0.1, 95% CI 2-sided [-5.2 to 5.5]

2. Secondary Outcome: Percentage of Participants With Favorable Clinical Response
Description: Percentage of participants who have no signs or symptoms of infection at the surgical site and do not require surgical intervention for infection
Time Frame: 4 weeks posttreatment
Population: Population analyzed was participants who had no signs or symptoms of infection at the surgical site and did not require surgical intervention for infection.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ertapenem | Ceftriaxone/Metronidazole
Number analyzed (Participants) | 251 | 248
percentage of participants | 96.8 [94.6 to 99.0] | 95.5 [93.0 to 98.1]
Statistical Analysis 1: Comparison: Ertapenem vs Ceftriaxone/Metronidazole; Test type: Superiority or Other; Miettinen and Nurminen; Difference in percentage of prophylaxis = 1.3, 95% CI 2-sided [-2.2 to 5.1]

ADVERSE EVENTS:
Time Frame: Up to and including 28 days after last administration of study drug
Arm/Group | Ertapenem | Ceftriaxone/Metronidazole
Serious Adverse Events (participants affected / at risk) | 6/290 | 14/297
Other Adverse Events (participants affected / at risk) | 23/290 | 18/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertapenem (N=290) | Ceftriaxone/Metronidazole (N=297)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Incision Site Infection (Infections and infestations) | 0 (0) | 1 (1)
Pelvic Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic Fistula (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anastomotic Leak (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Vocal Cord Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Embolism Venous (Vascular disorders) | 0 (0) | 1 (1)
Venous Thrombosis Limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertapenem (N=290) | Ceftriaxone/Metronidazole (N=297)
Pyrexia (General disorders) | 23 (24) | 18 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.